CLINICAL TRIAL: NCT01844986
Title: A Phase III, Randomised, Double Blind, Placebo Controlled, Multicentre Study of Olaparib Maintenance Monotherapy in Patients With BRCA Mutated Advanced (FIGO Stage III-IV) Ovarian Cancer Following First Line Platinum Based Chemotherapy.
Brief Title: Olaparib Maintenance Monotherapy in Patients With BRCA Mutated Ovarian Cancer Following First Line Platinum Based Chemotherapy.
Acronym: SOLO-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: GOG Foundation (Network); Myriad Genetic Laboratories, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0818C00001; 2024-511142-39-00 (Registry Identifier: CTIS (EU)); 2013-001551-13 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Newly Diagnosed; Advanced Ovarian Cancer; FIGO Stage III-IV; BRCA Mutation; Complete Response; Partial Response; First Line Platinum Chemotherapy
Keywords: BRCA; Ovarian Cancer; Chemotherapy; PARP inhibitor; First Line; FIGO Stage III; FIGO Stage IV
MeSH Terms: conditions — Pathologic Complete Response; Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib tablets p.o. 300mg twice daily (Experimental): Olaparib/placebo tablets p.o 300mg twice daily for up to 3 years or until objective radiological disease progression as per RECIST as assessed by the Investigator. Patients with evidence of stable disease (or those who have progressed), may continue on treatment beyond 2 years, if in the patient's best interest. Dose reduction to 250mg and subsequently 200mg is permitted following confirmation of toxicity
  Interventions: Drug: Olaparib 300mg tablets
- Placebo tablets p.o. twice daily (Placebo Comparator): Olaparib/placebo tablets p.o 300mg twice daily for up to 3 years or until objective radiological disease progression as per RECIST as assessed by the Investigator. Patients with evidence of stable disease (or those who have progressed), may continue on treatment beyond 2 years, if in the patient's best interest. Dose reduction to 250mg and subsequently 200mg is permitted following confirmation of toxicity
  Interventions: Drug: Olaparib 300mg tablets

INTERVENTIONS:
Drug: Olaparib 300mg tablets — Olaparib/placebo tablets p.o 300mg twice daily for up to 2 years or until objective radiological disease progression as per RECIST as assessed by the Investigator. Patients with evidence of stable disease (or those who have progressed), may continue on treatment beyond 2 years, if in the patient's best interest. Dose reduction to 250mg and subsequently 200mg is permitted following confirmation of toxicity.

SUMMARY:
Olaparib Monotherapy in Patients with BRCA Mutated Ovarian Cancer following First Line Platinum Based Chemotherapy.

DETAILED DESCRIPTION:
A Phase III, Randomised, Double Blind, Placebo Controlled, Multicentre Study of Olaparib Maintenance Monotherapy in Patients with BRCA Mutated Advanced (FIGO Stage III-IV) Ovarian Cancer following First Line Platinum Based Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with newly diagnosed, histologically confirmed, high risk advanced (FIGO stage III - IV) BRCA mutated high grade serous or high grade endometrioid ovarian cancer, primary peritoneal cancer and / or fallopian - tube cancer who have completed first line platinum based chemotherapy (intravenous or intraperitoneal).
* Stage III patients must have had one attempt at optimal debulking surgery (upfront or interval debulking). Stage IV patients must have had either a biopsy and/or upfront or interval debulking surgery.
* Documented mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function).
* Patients who have completed first line platinum (e.g. carboplatin or cisplatin), containing therapy (intravenous or intraperitoneal) prior to randomisation:
* Patients must have, in the opinion of the investigator, clinical complete response or partial response and have no clinical evidence of disease progression on the post treatment scan or rising CA-125 level, following completion of this chemotherapy course. Patients with stable disease on the post-treatment scan at completion of first line platinum-containing therapy are not eligible for the study.
* Patients must be randomized within 8 weeks of their last dose of chemotherapy

Exclusion Criteria:

* BRCA1 and/or BRCA2 mutations that are considered to be non detrimental (e.g. "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favor polymorphism" or "benign polymorphism" etc).
* Patients with early stage disease (FIGO Stage I, IIA, IIB or IIC)
* Stable disease or progressive disease on the post-treatment scan or clinical evidence of progression at the end of the patient's first line chemotherapy treatment.
* Patients where more than one debulking surgery has been performed before randomisation to the study. (Patients who, at the time of diagnosis, are deemed to be unresectable and undergo only a biopsy or oophorectomy but then go on to receive chemotherapy and interval debulking surgery are eligible).
* Patients who have previously been diagnosed and treated for earlier stage ovarian, fallopian tube or primary peritoneal cancer.
* Patients who have previously received chemotherapy for any abdominal or pelvic tumour, including treatment for prior diagnosis at an earlier stage for their ovarian, fallopian tube or primary peritoneal cancer. (Patients who have received prior adjuvant chemotherapy for localised breast cancer may be eligible, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease).
* Patients with synchronous primary endometrial cancer unless both of the following criteria are met: 1) stage <2 2) less than 60 years old at the time of diagnosis of endometrial cancer with stage IA or IB grade 1 or 2, or stage IA grade 3 endometrioid adenocarcinoma OR ≥ 60 years old at the time of diagnosis of endometrial cancer with Stage IA grade 1 or 2 endometrioid adenocarcinoma. Patients with serous or clear cell adenocarcinoma or carcinosarcoma of the endometrium are not eligible.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-08-26 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2028-08-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Paul DiSilvestro, MD, Principal Investigator — Women & Infants Hospital, Providence, Rhode Island, USA; Prof Kathleen Moore, MD, Principal Investigator — University of Oklahoma Health Sciences Center, Oklahoma City, USA
Locations (177):
- United States (81):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Kaiser Permanente, Oakland, California
  - Kaiser Permanente, Roseville, California
  - Stanford Women's Cancer Center, Stanford, California
  - Babak Edraki, Walnut Creek, California
  - University of Colorado, Aurora, Colorado
  - Univ of Connecticut Health Center, Farmington, Connecticut
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Gynecologic Cancer Center, Orlando, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Nancy N. & J.C. Lewis Cancer and Research Pavillion, Savannah, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Univ Chicago Medical Center, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Vincent Hospital & Health Care Center, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, Mishawaka, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Norton Cancer Institute Research, Louisville, Kentucky
  - Maine Medical Partners, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Gynecologic Oncology of West MI, PLLC, Grand Rapids, Michigan
  - Minnesota Oncology Hematology, PA, Edina, Minnesota
  - Mayo Clinic - Rochester, MN, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Valley Cancer Consortium CCOP, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Womens Cancer Center of Nevada, Las Vegas, Nevada
  - MD Anderson at Cooper Cancer Center, Camden, New Jersey
  - John Theurer Cancer Center, Hackensack, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Women's Cancer Care Associates, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai Medical Center - New York, New York, New York
  - Perlmutter Cancer Center, New York, New York
  - Hope Women's Cancer Centers, Asheville, North Carolina
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Hospital, Canton, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Clinic Women's Health, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center of Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Aurora Baycare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Froedtert Memorial Hospital, Milwaukee, Wisconsin
- Australia (3):
  - Mercy Hospital for Women, Heidelberg
  - The Royal Womens Hospital, Parkville
  - Prince of Wales Hospital, Randwick
- Brazil (8):
  - Centro Diagnóstico Barretos, Barretos
  - Hospital Araujo Jorge, Goiânia
  - Centro de Novos Tratamentos Itajai, Itajaí
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericordia de Porto Alagre, Porto Alegre
  - Hospital de Base São José do Rio Preto, São José do Rio Preto
  - Centro de Referencia da Saude da Mulher, São Paulo
  - Instituto do Câncer de São Paulo, São Paulo
- Canada (7):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - CHUM - Hopital Norte-Dame, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
- China (16):
  - Beijing Cancer Hospital, Beijing
  - The Tumor Hospital affiliated to China Medical Science Insti, Beijing
  - 1st Hospital of Jilin university, Changchun
  - Jilin Provincial Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital Affiliated to Sichuan University, Chengdu
  - ChongQing Cancer Hospital, Chongqing
  - Research Site, Guangzhou
  - Women's Hospital, Zhejaing University School of Medicine, Hangzhou
  - The Tumour Hospital of Harbin Medical University, Harbin
  - Zhejiang Cancer Hospital, Huangzhou, Huangzhou
  - JINAN, Qi Lu Hosp. of SD Univ., Jinan
  - Obstetris and Gynecology Hospital of Fudan University, Shanghai
  - Shanghai Cancer Hospital of Fudan University, Shanghai
  - The First Affiliated Hospital of Soochow Universit, Suzhou
  - First affiliated hospital college of XianJiaotong University, Xi'an
- France (7):
  - Institut Bergonie, Bordeaux
  - CAC François Baclesse, Caen
  - 69LYON, C Bérard, Onco, Lyon
  - Centre Catherine de Sienne, Nantes
  - 75PARIS, H Tenon, Onco, Paris
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Sapir Medical Centre, Kfar Saba
  - Rabin MC, Petah Tikva
  - Tel-Aviv Sourkasy Medical Center, Tel Aviv
  - Chaim Sheba Medical Centre, Tel Litwinsky
- Italy (8):
  - Bari- Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliera "Cannizzaro", Catania
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Per Cura Tumori - Milano, Milan
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto Irccs, Padua
  - Istituto Regina Elena-Polo Oncologico Ifo, Roma
  - Policlinico Universitario A. Gemelli, Roma
- Japan (8):
  - Hyogo CC, Akashi-shi
  - National Cancer Center Hosp, Chūōku
  - NHO Kyushu CC, Fukuoka
  - Saitama Med. Univ. Int. Med. C, Hidaka-shi
  - NHO Shikoku Cancer Center, Matsuyama
  - Niigata Univ. Med. Dent., Niigata
  - Hokkaido University Hospital, Sapporo
  - Shizuoka Cancer Center, Sunto-gun
- Netherlands (2):
  - Netherlands Cancer Institute Antoni van Leeuwenhoek Hospital, Amsterdam
  - Maastricht Universitair Medisch Centrum, Maastricht
- Poland (5):
  - Niepubliczny Zaklad Opieki Zdrowotnej Innowacyjna Medycyna, Grzepnica
  - SPZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii, Olsztyn
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Szpital Specjalistyczny im. Swietej Rodziny SPZOZ, Warsaw
- Russia (7):
  - Udmurtia Republic Clinical Oncology Center, Izhevsk
  - Chemotherapy Department, Russian Cancer Research Centre, Moscow
  - State Institution of Heath Omsk Regional Oncology Dispensary, Omsk
  - Cancer Research Institute, Saint Petersburg
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - St.Petersburg City Oncology Dispensary, Dept. Gynecology, Saint Petersburg
  - Research Institute of Oncology RAMS, Tomsk
- South Korea (6):
  - National Cancer Center, Goyang-si
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (7):
  - Barcelona,H.Vall d´Hebrón,Oncología, Barcelona
  - Córdoba,H.Reina Sofía,Oncología, Córdoba
  - H.Llobregat,ICO-Duran i Reynals,Oncología, Hospitalet deLlobregat(Barcelo
  - Madrid, MD Anderson, Oncología, Madrid
  - Madrid,H.U.La Paz,Oncología, Madrid
  - Valencia, IVO, Oncología, Valencia
  - Valencia,H.C.U.Valencia,Oncología, Valencia
- United Kingdom (7):
  - City Hospital, Birmingham, Cancer Trials Team, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Arden Cancer Centre, Coventry
  - Edinburgh Cancer Research UK Centre, Edinburgh
  - Cancer Research UK and UCL Cancer Trials Centre, London
  - Royal Marsden Hospital, London
  - Royal Marsden Hospital and Institute of Cancer Research, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Barnicle A, Ray-Coquard I, Rouleau E, Cadoo K, Simpkins F, Aghajanian C, Leary A, Poveda A, Lheureux S, Pujade-Lauraine E, You B, Ledermann J, Matulonis U, Gourley C, Timms KM, Lai Z, Hodgson DR, Elks CE, Dearden S, Egile C, Lao-Sirieix P, Harrington EA, Brown JS. Patterns of genomic instability in > 2000 patients with ovarian cancer across six clinical trials evaluating olaparib. Genome Med. 2024 Dec 18;16(1):145. doi: 10.1186/s13073-024-01413-5. PMID 39695768
- [Derived] DiSilvestro P, Banerjee S, Colombo N, Scambia G, Kim BG, Oaknin A, Friedlander M, Lisyanskaya A, Floquet A, Leary A, Sonke GS, Gourley C, Oza A, Gonzalez-Martin A, Aghajanian C, Bradley W, Mathews C, Liu J, McNamara J, Lowe ES, Ah-See ML, Moore KN; SOLO1 Investigators. Overall Survival With Maintenance Olaparib at a 7-Year Follow-Up in Patients With Newly Diagnosed Advanced Ovarian Cancer and a BRCA Mutation: The SOLO1/GOG 3004 Trial. J Clin Oncol. 2023 Jan 20;41(3):609-617. doi: 10.1200/JCO.22.01549. Epub 2022 Sep 9. PMID 36082969
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Banerjee S, Moore KN, Colombo N, Scambia G, Kim BG, Oaknin A, Friedlander M, Lisyanskaya A, Floquet A, Leary A, Sonke GS, Gourley C, Oza A, Gonzalez-Martin A, Aghajanian C, Bradley WH, Holmes E, Lowe ES, DiSilvestro P. Maintenance olaparib for patients with newly diagnosed advanced ovarian cancer and a BRCA mutation (SOLO1/GOG 3004): 5-year follow-up of a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2021 Dec;22(12):1721-1731. doi: 10.1016/S1470-2045(21)00531-3. Epub 2021 Oct 26. PMID 34715071
- [Derived] Friedlander M, Moore KN, Colombo N, Scambia G, Kim BG, Oaknin A, Lisyanskaya A, Sonke GS, Gourley C, Banerjee S, Oza A, Gonzalez-Martin A, Aghajanian C, Bradley WH, Liu J, Mathews C, Selle F, Lortholary A, Lowe ES, Hettle R, Flood E, Parkhomenko E, DiSilvestro P. Patient-centred outcomes and effect of disease progression on health status in patients with newly diagnosed advanced ovarian cancer and a BRCA mutation receiving maintenance olaparib or placebo (SOLO1): a randomised, phase 3 trial. Lancet Oncol. 2021 May;22(5):632-642. doi: 10.1016/S1470-2045(21)00098-X. Epub 2021 Apr 13. PMID 33862001
- [Derived] Moore K, Colombo N, Scambia G, Kim BG, Oaknin A, Friedlander M, Lisyanskaya A, Floquet A, Leary A, Sonke GS, Gourley C, Banerjee S, Oza A, Gonzalez-Martin A, Aghajanian C, Bradley W, Mathews C, Liu J, Lowe ES, Bloomfield R, DiSilvestro P. Maintenance Olaparib in Patients with Newly Diagnosed Advanced Ovarian Cancer. N Engl J Med. 2018 Dec 27;379(26):2495-2505. doi: 10.1056/NEJMoa1810858. Epub 2018 Oct 21. PMID 30345884
- See also: Redacted Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1817&filename=SOLO1_Clinical%20Study%20Protocol.pdf
- See also: Redacted Statistical Analysis Plan — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1817&filename=SOLO1_Statistical%20Analysis%20Plan.pdf
- See also: Redacted Statistical Analysis Plan — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1817&filename=SOLO1_Statistiacal%20Analysis%20Plan..pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Global Cohort: 391 randomised. First/Last patient randomised 03Sep2013/06Mar2015.
  China Cohort: 64 randomised. First/Last patient randomised 09Jan2015/22Mar2016.
  A total of 450 patients randomised (386 global cohort only, 64 China cohort (of which 5 included in global cohort)). Global Cohort used for hypotheses testing of study.
Pre-assignment Details: It was planned that approximately 344 women in the Global Cohort, and 53 women in the China Cohort, with BRCA mutated ovarian cancer patients who are in clinical complete or partial response following first line platinum based chemotherapy were to receive olaparib 300 mg bd or matching placebo in a 2:1 ratio.
Groups:
- Olaparib 300mg Tablets; Placebo Tablets: Taken orally twice daily
Period: Overall Study (Global Cohort)
Arm/Group | Olaparib 300mg Tablets | Placebo Tablets
Started ((Randomised to study treatment)) | 260 | 131
Completed ((Ongoing study at time of PFS analysis DCO:17 May 2018)) | 183 | 91
Not Completed | 77 | 40
Not completed — Severe non-compliance to protocol | 1 | 0
Not completed — Withdrawal by Subject | 21 | 14
Not completed — Death | 55 | 26
Period: Overall Study (China Cohort)
Arm/Group | Olaparib 300mg Tablets | Placebo Tablets
Started ((Randomised to study treatment)) | 44 | 20
Completed ((Ongoing study at time of PFS analysis DCO:17 May 2018)) | 33 | 14
Not Completed | 11 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 10 | 6

BASELINE CHARACTERISTICS:
Population: Global Cohort (391 subjects):
  260 Olaparib 131 Placebo
  China Cohort (64 subjects):
  44 Olaparib 20 Placebo
  Included in both cohorts (5 subjects):
  4 Olaparib
  1 Placebo
  Total (450 subjects):
  300 Olaparib 150 Placebo
Groups:
- Olaparib 300mg Tablets (Global Cohort & China Cohort); Placebo Tablets (Global Cohort & China Cohort): Taken orally twice daily
- Total: Total of all reporting groups
Arm/Group | Olaparib 300mg Tablets (Global Cohort & China Cohort) | Placebo Tablets (Global Cohort & China Cohort) | Total
Number analyzed (Participants) | 300 | 150 | 450
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Each study is reported in a separate row. There were 4 participants who were in both the Global and China Olaparib Arm, and 1 participant in both the Global and China Placebo Arm.
  Years
    Global Cohort: number analyzed (Participants) | 260 | 131 | 391
    Global Cohort | 53.6 (9.38) | 53.4 (9.79) | 53.5 (9.51)
    China Cohort: number analyzed (Participants) | 44 | 20 | 64
    China Cohort | 50.7 (7.27) | 51.5 (7.95) | 51.0 (7.44)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each study is reported in a separate row. There were 4 participants who were in both the Global and China Olaparib Arm, and 1 participant in both the Global and China Placebo Arm.
  Participants
    Global Cohort: number analyzed (Participants) | 260 | 131 | 391
    Global Cohort: Female | 260 | 131 | 391
    Global Cohort: Male | 0 | 0 | 0
    China Cohort: number analyzed (Participants) | 44 | 20 | 64
    China Cohort: Female | 44 | 20 | 64
    China Cohort: Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each study is reported in a separate row. There were 4 participants who were in both the Global and China Olaparib Arm, and 1 participant in both the Global and China Placebo Arm.
  Participants
    Global Cohort: number analyzed (Participants) | 260 | 131 | 391
    Global Cohort: American Indian or Alaska Native | 0 | 1 | 1
    Global Cohort: Asian | 39 | 20 | 59
    Global Cohort: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Global Cohort: Black or African American | 2 | 2 | 4
    Global Cohort: White | 214 | 106 | 320
    Global Cohort: More than one race | 1 | 0 | 1
    Global Cohort: Unknown or Not Reported | 3 | 1 | 4
    China Cohort: number analyzed (Participants) | 44 | 20 | 64
    China Cohort: American Indian or Alaska Native | 0 | 0 | 0
    China Cohort: Asian | 44 | 20 | 64
    China Cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    China Cohort: Black or African American | 0 | 0 | 0
    China Cohort: White | 0 | 0 | 0
    China Cohort: More than one race | 0 | 0 | 0
    China Cohort: Unknown or Not Reported | 0 | 0 | 0
Response to previous platinum chemotherapy (as randomised) [Count of Participants; unit: Participants] — Population: Each study is reported in a separate row. There were 4 participants who were in both the Global and China Olaparib Arm, and 1 participant in both the Global and China Placebo Arm.
  Participants
    Global Cohort: number analyzed (Participants) | 260 | 131 | 391
    Global Cohort: Complete Response | 213 | 107 | 320
    Global Cohort: Partial Response | 47 | 24 | 71
    China Cohort: number analyzed (Participants) | 44 | 20 | 64
    China Cohort: Complete Response | 37 | 18 | 55
    China Cohort: Partial Response | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Using Investigator Assessment According to Modified Response Evaluation Criteria in Solid Tumours (RECIST 1.1)
Description: To determine the efficacy by progression free survival (PFS) using investigator assessment according to modified Response Evaluation Criteria in Solid Tumours (RECIST 1.1) of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy.
Time Frame: Radiologic scans performed at baseline then every 12 weeks up to 156 weeks, then every 24 weeks thereafter until objective radiological disease progression. DCO: 17 May 2018
Population: Global Full Analysis Set (FAS) consisting of all patients randomized as part of global recruitment (including 5 patients randomized in China) [Primary analysis] China Full Analysis Set (FAS) consisting of all patients randomized at sites in China (including 5 patients also included in the Global Cohort).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Olaparib 300mg Tablets (Global Cohort); Placebo Tablets (Global Cohort); Olaparib 300mg Tablets (China Cohort); Placebo Tablets (China Cohort): Taken orally twice daily
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 260 | 131 | 44 | 20
Months | NA [NA to NA] — Insufficient PFS events to estimate median, lower and upper confidence limit. | 13.8 [11.1 to 18.2] | NA [NA to NA] — Insufficient PFS events to estimate median, lower and upper confidence limit. | 9.3 [6.4 to NA] — Insufficient PFS events to estimate upper confidence limit.
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p < 0.0001, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy; Model includes a factor for response to previous platinum chemotherapy; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.23 to 0.41] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes the stratification variable of response to first-line platinum chemotherapy as a covariate; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.23 to 0.97] — A hazard ratio < 1 favours olaparib

2. Secondary Outcome: Efficacy in Patients Following First Line Platinum Based Chemotherapy by Assessment of Overall Survival
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of overall survival (OS). Reports results of a pre-specified interim analysis; results for final OS analysis (235 OS events) anticipated 2029.
Time Frame: Assessed every 4 weeks until treatment discontinues (up to a max of 156 weeks), then as per protocol. Analysis performed with DCO: 17May2018. Further analyses will be performed at 7 years (descriptive), after 206 events and after 60% maturity.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 260 | 131 | 44 | 20
Months | NA [NA to NA] — Insufficient OS events to estimate median, lower and upper confidence limit. | NA [NA to NA] — Insufficient OS events to estimate median, lower and upper confidence limit. | NA [NA to NA] — Insufficient OS events to estimate median, lower and upper confidence limit. | NA [NA to NA] — Insufficient OS events to estimate median, lower and upper confidence limit.
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p = 0.8903, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy; Model includes a factor for response to previous platinum chemotherapy; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.60 to 1.53] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes the stratification variable of response to first-line platinum chemotherapy as a covariate; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.29 to 2.28] — A hazard ratio < 1 favours olaparib

3. Secondary Outcome: Efficacy in Patients Following First Line Platinum Based Chemotherapy by Assessment of Time to Earliest Progression by RECIST or Cancer Antigen (CA-125) or Death
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of time to earliest progression by RECIST or Cancer Antigen-125 (CA-125) or death
Time Frame: CA-125 performed at baseline + every 4 weeks. Radiologic scans performed at baseline + every 12 weeks up to 156 weeks, then every 24 weeks until objective radiological disease progression. DCO:17May2018
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 260 | 131 | 44 | 20
Months | NA [NA to NA] — Insufficient events to estimate median, lower and upper confidence limit. | 12.0 [10.8 to 16.6] | NA [NA to NA] — Insufficient events to estimate median, lower and upper confidence limit. | 8.9 [6.4 to NA] — Insufficient events to estimate upper confidence limit.
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p < 0.0001, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy; Model includes a factor for response to previous platinum chemotherapy; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.23 to 0.40] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority; Regression, Cox — Not applicable due to small sample size. China cohort designed to provide descriptive analysis only; Model includes the stratification variable of response to first-line platinum chemotherapy as a covariate; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.23 to 0.99] — A hazard ratio <1 favours Olaparib

4. Secondary Outcome: Efficacy in Patients Following First Line Platinum Based Chemotherapy by Assessment of Time From Randomization to Second Progression
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of time from randomisation to second progression (PFS2)
Time Frame: Following first progression disease then assessed per local practice every 12 weeks until second progression.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 260 | 131 | 44 | 20
Months | NA [NA to NA] — Insufficient PFS2 events to estimate median, lower and upper confidence limit. | 41.9 [36.5 to 47.9] | NA [NA to NA] — Insufficient PFS2 events to estimate median, lower and upper confidence limit. | NA [NA to NA] — Insufficient PFS2 events to estimate median, lower and upper confidence limit.
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p = 0.0002, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy; Model includes a factor for response to previous platinum chemotherapy; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.35 to 0.72] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes the stratification variable of response to first-line platinum chemotherapy as a covariate; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.23 to 1.35] — A hazard ratio <1 favours Olaparib

5. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) as Assessed by the the Trial Outcome Index (TOI) of the Functional Assessment of Cancer Therapy - Ovarian (FACT-O)
Description: To compare the effects of olaparib maintenance monotherapy compared to placebo on Health-related Quality of Life (HRQoL) as assessed by the trial outcome index (TOI) of the Functional Assessment of Cancer Therapy - Ovarian (FACT-O) in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy. The TOI ranges from 0-100 and a higher score indicates a higher HRQoL.
Time Frame: Questionnaires will be given to the patient at baseline, at Day 29 and then every 12 weeks for 156 weeks, then every 24 weeks or until the data cut off for the PFS analysis, change in TOI over 24 months reported
Population: Global Full Analysis Set (FAS) consisting of all patients randomized as part of global recruitment (including 5 patients randomized in China) with a baseline and post baseline TOI scores available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort)
Number analyzed (Participants) | 260 | 131
Scores on a scale | 0.30 [-0.717 to 1.318] | 3.30 [1.839 to 4.758]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p = 0.0010, Mixed Models Analysis; Fixed effects for treatment, visit and baseline TOI with the treatment by visit and baseline TOI by visit interaction. Random patient effect; Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-4.779 to -1.216]

6. Secondary Outcome: Efficacy in Patients Following First Line Platinum Based Chemotherapy by Assessment of Time to First Subsequent Therapy or Death (TFST)
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of time from randomisation to first subsequent therapy or death (TFST). Reports results of a pre-specified interim analysis; final analysis results will later be added at time of final OS analysis (anticipated 2029).
Time Frame: Assessed every 12 weeks following treatment discontinuation. Analysis performed with DCO: 17May2018. Further analyses will be performed at 7 years (descriptive), after 206 events and after 60% maturity.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 260 | 131 | 44 | 20
Months | 51.8 [44.3 to NA] — Insufficient events to estimate upper confidence limit. | 15.1 [12.7 to 20.5] | 34.3 [23.1 to NA] — Insufficient events to estimate upper confidence limit. | 10.3 [6.9 to NA] — Insufficient events to estimate upper confidence limit.
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p < 0.0001, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy; Model includes a factor for response to previous platinum chemotherapy; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.22 to 0.40] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes the stratification variable of response to first-line platinum chemotherapy as a covariate; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.29 to 1.23] — A hazard ratio <1 favours Olaparib

7. Secondary Outcome: Efficacy in Patients Following First Line Platinum Based Chemotherapy by Assessment of Time to Second Subsequent Therapy or Death (TSST)
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of time from randomisation to second subsequent therapy or death (TSST). Reports results of a pre-specified interim analysis; final analysis results will later be added at time of final OS analysis (anticipated 2029).
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 260 | 131 | 44 | 20
Months | NA [NA to NA] — Insufficient events to estimate median, lower and upper confidence limit. | 40.7 [32.9 to 47.7] | NA [NA to NA] — Insufficient events to estimate median, lower and upper confidence limit. | 27.4 [19.4 to NA] — Insufficient events to estimate upper confidence limit.
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p < 0.0001, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy; Model includes a factor for response to previous platinum chemotherapy; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.32 to 0.63] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes the stratification variable of response to first-line platinum chemotherapy as a covariate; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.25 to 1.26] — A hazard ratio <1 favours Olaparib

8. Secondary Outcome: Efficacy in Patients Following First Line Platinum Based Chemotherapy by Assessment of Time From Randomization to Study Treatment Discontinuation or Death (TDT)
Description: To determine the efficacy of olaparib maintenance monotherapy compared to placebo in BRCA mutated high risk advanced ovarian cancer patients who are in clinical complete response or partial response following first line platinum based chemotherapy by assessment of time from randomisation to study treatment discontinuation or death (TDT). Reports results of a pre-specified interim analysis; final analysis results will later be added at time of final OS analysis (anticipated 2029).
Time Frame: Time elapsed from randomization to study treatment discontinuation or death. Analysis performed with DCO: 17May2018. Further analyses will be performed at 7 years (descriptive), after 206 events and after 60% maturity.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
Number analyzed (Participants) | 260 | 131 | 44 | 20
Months | 24.6 [24.0 to 24.8] | 13.8 [11.2 to 16.4] | 24.8 [14.2 to 24.9] | 8.6 [5.9 to 24.8]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p < 0.0001, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy; Model includes a factor for response to previous platinum chemotherapy; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.51 to 0.79] — A hazard ratio < 1 favours olaparib
Statistical Analysis 2: Comparison: Olaparib 300mg Tablets (China Cohort) vs Placebo Tablets (China Cohort); Test type: Superiority; Regression, Cox — Not applicable, due to small sample size. China cohort designed to provide descriptive analysis only; Model includes the stratification variable of response to first-line platinum chemotherapy as a covariate; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.47 to 1.42] — A hazard ratio <1 favours Olaparib

9. Secondary Outcome: Efficacy in Patients With a Deleterious or Suspected Deleterious Variant in Either of the BRCA Genes by Assessment of PFS
Description: To assess efficacy of olaparib in patients identified as having a deleterious or suspected deleterious variant in either of the BRCA genes using variants identified with current and potential future BRCA mutation assays (gene sequencing and large rearrangement analysis)
Time Frame: Radiologic scans performed at baseline then every 12 weeks for the first 156 weeks, then every 24 weeks thereafter, assessed until disease progression. Analysis of data assessed up to a maximum of 54 months.
Population: Global Full Analysis Set (FAS) consisting of all patients randomized as part of global recruitment (including 5 patients randomized in China) and confirmed as Myriad gBRCAm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort)
Number analyzed (Participants) | 253 | 130
Months | NA [NA to NA] — Insufficient PFS events to estimate median, lower and upper confidence limit. | 13.8 [11.1 to 18.2]
Statistical Analysis 1: Comparison: Olaparib 300mg Tablets (Global Cohort) vs Placebo Tablets (Global Cohort); Test type: Superiority; p < 0.0001, Regression, Cox — Determined using a log-rank test stratified by response to previous platinum chemotherapy; Model includes a factor for response to previous platinum chemotherapy; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.22 to 0.40] — A hazard ratio < 1 favours olaparib

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from informed consent through treatment and safety follow-up period (30 days after study drug discontinued). Global cohort subjects were treated for an average of 1.7 years in Olaparib arm and 1.3 years in placebo arm. Subjects were followed up for all-cause mortality to end of study (no pre-specified max time). Global cohort subjects without a death reported were followed up for an average of 43.5 months in Olaparib arm and 42.5 months in placebo arm.
Description: Adverse events summaries showing subjects at risk are based on those subjects who received treatment. The summary of All cause mortality showing subjects at risk are based on those subjects who are randomised (irrespective of whether received treatment or not). Note 1 subject in Global cohort placebo arm was randomised but not treated.
Arm/Group | Olaparib 300mg Tablets (Global Cohort) | Placebo Tablets (Global Cohort) | Olaparib 300mg Tablets (China Cohort) | Placebo Tablets (China Cohort)
All-Cause Mortality (participants affected / at risk) | 55/260 | 27/131 | 10/44 | 6/20
Serious Adverse Events (participants affected / at risk) | 54/260 | 16/130 | 13/44 | 3/20
Other Adverse Events (participants affected / at risk) | 253/260 | 117/130 | 43/44 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300mg Tablets (Global Cohort) (N=260) | Placebo Tablets (Global Cohort) (N=130) | Olaparib 300mg Tablets (China Cohort) (N=44) | Placebo Tablets (China Cohort) (N=20)
Anaemia (Blood and lymphatic system disorders) | 17 (36) | 0 (0) | 8 (10) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic cyst (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300mg Tablets (Global Cohort) (N=260) | Placebo Tablets (Global Cohort) (N=130) | Olaparib 300mg Tablets (China Cohort) (N=44) | Placebo Tablets (China Cohort) (N=20)
Anaemia (Blood and lymphatic system disorders) | 90 (156) | 12 (18) | 21 (44) | 3 (3)
Palpitations (Cardiac disorders) | 12 (19) | 2 (2) | 3 (6) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 8 (10) | 2 (3) | 5 (8) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 18 (22) | 10 (10) | 2 (3) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 63 (86) | 25 (28) | 2 (4) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 8 (8) | 4 (4) | 1 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 43 (50) | 16 (18) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 201 (412) | 49 (75) | 28 (49) | 5 (11)
Stomatitis (Gastrointestinal disorders) | 23 (37) | 3 (5) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 8 (8) | 4 (4) | 3 (3) | 2 (2)
Fatigue (General disorders) | 106 (138) | 39 (48) | 16 (22) | 3 (3)
Influenza like illness (General disorders) | 19 (29) | 11 (11) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 24 (32) | 9 (10) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 15 (19) | 5 (8) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 28 (36) | 12 (15) | 17 (20) | 6 (13)
Alanine aminotransferase increased (Investigations) | 9 (13) | 8 (8) | 6 (23) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 11 (13) | 6 (7) | 6 (15) | 3 (6)
Blood creatinine increased (Investigations) | 21 (30) | 2 (4) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (17) | 10 (15) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 66 (88) | 35 (47) | 2 (2) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (50) | 16 (22) | 3 (6) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (36) | 13 (17) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (34) | 11 (15) | 1 (4) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 16 (33) | 5 (5) | 15 (64) | 2 (6)
Neutropenia (Blood and lymphatic system disorders) | 40 (84) | 9 (11) | 17 (68) | 1 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (52) | 2 (4) | 13 (35) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 46 (61) | 17 (22) | 9 (14) | 0 (0)
Constipation (Gastrointestinal disorders) | 72 (97) | 25 (30) | 8 (10) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 89 (205) | 32 (58) | 8 (12) | 4 (10)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Mouth ulceration (Gastrointestinal disorders) | 5 (11) | 0 (0) | 5 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 104 (242) | 19 (26) | 18 (38) | 3 (4)
Asthenia (General disorders) | 63 (131) | 16 (20) | 3 (6) | 1 (2)
Mucosal inflammation (General disorders) | 17 (27) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 31 (40) | 12 (15) | 8 (8) | 2 (2)
Influenza (Infections and infestations) | 19 (24) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 27 (38) | 17 (37) | 5 (16) | 3 (15)
Pharyngitis (Infections and infestations) | 9 (11) | 3 (6) | 4 (5) | 0 (0)
Sinusitis (Infections and infestations) | 11 (12) | 8 (8) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 29 (52) | 8 (10) | 4 (4) | 2 (2)
Neutrophil count decreased (Investigations) | 20 (40) | 7 (14) | 7 (17) | 2 (6)
Platelet count decreased (Investigations) | 8 (12) | 2 (4) | 6 (19) | 0 (0)
Weight increased (Investigations) | 13 (15) | 12 (12) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 16 (37) | 6 (9) | 10 (28) | 2 (9)
Decreased appetite (Metabolism and nutrition disorders) | 51 (68) | 13 (19) | 17 (22) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (24) | 3 (6) | 3 (10) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 (22) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 11 (13) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 51 (68) | 20 (23) | 8 (10) | 6 (16)
Dysgeusia (Nervous system disorders) | 68 (92) | 5 (6) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 58 (109) | 30 (40) | 7 (9) | 3 (10)
Hypoaesthesia (Nervous system disorders) | 5 (6) | 2 (3) | 4 (4) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 15 (15) | 7 (9) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 15 (15) | 11 (11) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 12 (14) | 13 (15) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 27 (31) | 16 (20) | 3 (3) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (57) | 28 (37) | 5 (6) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 (53) | 7 (7) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 12 (15) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 16 (23) | 11 (11) | 2 (4) | 1 (1)
Hot flush (Vascular disorders) | 17 (25) | 11 (12) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 9 (18) | 12 (17) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The data presented based on the March DCO (17 May 2018) are not the final analyses for OS, TFST, TSST, and TDT. Further analyses of these (numbered as endpoints 2, 6, 7 and 8 in Outcome Measures section) will be performed as planned in the protocol and SAP when the pre-specified number of OS events are achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT01844986/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT01844986/SAP_003.pdf